CLINICAL TRIAL: NCT03118453
Title: A Behavioural Medicine Approach in Physical Therapy for Treatment of Chronic Pain - Evaluation of the Implementation Process and Outcome
Brief Title: Implementation of a Behavioural Medicine Approach in Physical Therapy for Treatment of Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mälardalen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140369
Record Dates: First submitted 2017-03-20; First posted 2017-04-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: Musculoskeletal pain/*therapy; Behavioral medicine; Physical therapy; Cost-benefit analyses; Treatment outcome; Adults
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active implementation clinics (Experimental): Patients recruited by physical therapists who underwent an implementation period with active implementations strategies, such as supervision, web lectures, peer learning in groups consisting of colleagues. A behavioral medicine approach in physical therapy for patients with musculoskeletal pain was encouraged with these active implementation strategies.
  Interventions: Behavioral: Active implementation clinics
- Passive implementation clinics (Active Comparator): Patients recruited by physical therapists who underwent an implementation period with passive implementations strategies, such as written material and a short web lecture. A behavioral medicine approach in physical therapy for patients with musculoskeletal pain was encouraged with these passive implementation strategies
  Interventions: Behavioral: Passive implementation clinics

INTERVENTIONS:
Behavioral: Active implementation clinics — Physical therapy treatment as the physical therapist chooses
  Arms: Active implementation clinics
Behavioral: Passive implementation clinics — Physical therapy treatment as the physical therapist chooses
  Arms: Passive implementation clinics

SUMMARY:
Implementation of a behavioral medicine (BM) approach in physical therapy (PT) for patients with persistent musculoskeletal pain is in accordance with the state of science. Translation of research into clinical PT practice is challenging and may demand active implementation strategies.

The aim is to evaluate the implementation of a behavioural medicine approach for patients with persistent musculoskeletal pain concerning sustainable health benefits and sick-leave, as well as the cost-effectiveness of the implemented treatment.

Treatment outcomes for patients from two groups of physical therapists in primary care will be compared. In one group active implementation strategies have been employed, and in the other (control) passive implementation strategies during a 6-months intervention period. Patients are recruited during one-year after the implementation period.

The short and long-term effects of the implementation of the BM approach in PT treatment on patients' sick-leave, activity and participation, and health related quality of life will be compared to the patients from control condition clinics. The cost-effect and cost-benefit of an implementation of a behavioral medicine approach in physical therapy is evaluated from the perspective of the health care organization and society.

DETAILED DESCRIPTION:
The aim is to investigate the short and long-term effects for the implementation of a behavioral medicine approach in physical therapy on patients' sick-leave, activity and participation, and health related quality of life, compared to the control condition. Further the aim is to evaluate the cost-effect and cost-benefit of an active implementation of a behavioural medicine approach in physical therapy, compared to the passive implementation in the control condition.

In total 109 primary care patients with musculoskeletal pain ≥ 4 weeks are included consecutively in the active implementation and passive implementation (control) clinics. The sample size was based on a priori power analysis on differences in primary outcome between conditions and expected attrition. Patients from both conditions are included during the first year after the implementation period.

Data collection has been at onset and end of patients' treatment period, and will be at 6, 12, and 18 months post treatment (in both implementation and control clinics).

Recommended core outcomes regarding body structure, activity and participation are used. Primary outcomes: Participation in work life defined as days of sick-leave and participation in everyday life. Secondary outcomes will be patients' ratings of global treatment effects and pain intensity. Process measures: prognostic psychosocial factors possible to address in physical therapy such as functional self-efficacy, fear of movement and patient expectations on treatment effects. Depression, seen as a confounder, will be controlled for. Calculation of costs will include avoidable cost of the implementation, sunk costs will be ignored. Direct health care costs, i.e. use of health care services will be identified, measured and priced to assess costs from a societal perspective. Indirect costs, i.e. production loss due to sick leave and health care visits will be estimated. Cost-benefit will be calculated from the perspective of the society. Economic benefits will be measured as the net value of production gained for society, with an appropriate discount rate. Costs for society will be calculated on direct health care costs.

Data analyses: Regression models are used to compare patient outcomes between implementation and control clinics and performed per protocol and on an intention-to-treat-basis. Total costs, i.e. direct health care costs, direct and indirect non-health care costs and incremental costs, will be compared between conditions. A ratio between difference in outcome scores and costs between baseline and 6, 12, and 18 months post treatment will be. Incremental costs will be calculated per cost-benefit ratio associated with treatments in the two conditions. Bootstrapping is used for confidence intervals for cost-effectiveness and cost-benefit ratios.

ELIGIBILITY:
Inclusion criteria:

* Patients who presents for physical therapy in primary care.
* 18 - 65 years of age
* musculoskeletal pain for 4 weeks or more
* ability to speak and understand spoken and written Swedish

Exclusion criteria:

* systemic disease
* malignity
* serious spinal pathology
* osteoarthritis waiting for surgery
* diagnosed depression
* neurological disease or injury that severely affect activity capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-11; Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in days of sick-leave | through study completion, an average of 1 year
  Self-reports and sick-leave data from the Swedish Social Insurance Administration
Change in pain-related disability using Pain Disability Index | through study completion, an average of 1 year
  Pain Disability Index: Measure of disruptions in seven dimensions of everyday life. Self-reports on a11-graded numerical rating scale
Change in health related quality of life using EQ-5D | through study completion, an average of 1 year
  EuroQol, Quality of life scale in 5 dimensions (EQ-5D) which provides a simple descriptive profile and a single index value for health status.

SECONDARY OUTCOMES:
Change in the patients' perceptions of global treatment effect Change in perceived global treatment effect using the Patient Global Impression of Change Scale | through study completion, an average of 1 year
  Patients Global Impression of Change (PGIC) scale which provides the patient's belief about the treatment effect rated on a 7-graded scale
Change in self-efficacy for daily activities using the Self-efficacy Scale | through study completion, an average of 1 year
  The Self-efficacy Scale: ratings of self-efficacy for 20 common activities in daily life
Change in catastrophizing thoughts about pain using the Catastrophizing subscale of the Coping Strategies Questionnaire | through study completion, an average of 1 year
  The Catastrophizing subscale of the Coping Strategies Questionnaire: ratings of pain-related catastrophizing thoughts
Change in fear of movement/(re)injury using the Tampa Scale of Kinesiophobia | through study completion, an average of 1 year
  The Tampa Scale of Kinesiophobia: ratings of fear and avoidance of movement

CONTACTS AND LOCATIONS:
Overall Officials: Anne Söderlund, professor, Principal Investigator — Mälardalen University, Box 883, SE-721 23 Västerås, Sweden
Locations (3):
- Sweden (3):
  - Region Gävleborg, Gävle
  - Landstinget Sörmland, Nyköping
  - Region Västmanland, Västerås

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) because the participants have been assured of confidentiality and that only the researchers in the Project will have access to IPD

REFERENCES:
- [Background] Hill JC, Whitehurst DG, Lewis M, Bryan S, Dunn KM, Foster NE, Konstantinou K, Main CJ, Mason E, Somerville S, Sowden G, Vohora K, Hay EM. Comparison of stratified primary care management for low back pain with current best practice (STarT Back): a randomised controlled trial. Lancet. 2011 Oct 29;378(9802):1560-71. doi: 10.1016/S0140-6736(11)60937-9. Epub 2011 Sep 28. PMID 21963002
- [Background] Soderlund A, Lindberg P. Cognitive behavioural components in physiotherapy management of chronic whiplash associated disorders (WAD)--a randomised group study. G Ital Med Lav Ergon. 2007 Jan-Mar;29(1 Suppl A):A5-11. PMID 17650736
- [Background] Denison E, Asenlof P, Sandborgh M, Lindberg P. Musculoskeletal pain in primary health care: subgroups based on pain intensity, disability, self-efficacy, and fear-avoidance variables. J Pain. 2007 Jan;8(1):67-74. doi: 10.1016/j.jpain.2006.06.007. Epub 2006 Sep 1. PMID 16950657
- [Background] Asenlof P, Denison E, Lindberg P. Individually tailored treatment targeting activity, motor behavior, and cognition reduces pain-related disability: a randomized controlled trial in patients with musculoskeletal pain. J Pain. 2005 Sep;6(9):588-603. doi: 10.1016/j.jpain.2005.03.008. PMID 16139778
- [Background] Sandborgh M, Åsenlöf P, Lindberg P, Denison, E. Implementing behavioural medicine in physiotherapy treatment. Part II: Adherence to treatment protocol. Advances in Physiotherapy 12: 13-23, 2010 doi: 10.3109/14038190903480672
- [Background] Phillips CJ. Economic burden of chronic pain. Expert Rev Pharmacoecon Outcomes Res. 2006 Oct;6(5):591-601. doi: 10.1586/14737167.6.5.591. PMID 20528505
- [Background] Mantyselka PT, Kumpusalo EA, Ahonen RS, Takala JK. Direct and indirect costs of managing patients with musculoskeletal pain-challenge for health care. Eur J Pain. 2002;6(2):141-8. doi: 10.1053/eujp.2001.0311. PMID 11900474
- [Background] Lamb SE, Lall R, Hansen Z, Castelnuovo E, Withers EJ, Nichols V, Griffiths F, Potter R, Szczepura A, Underwood M; BeST trial group. A multicentred randomised controlled trial of a primary care-based cognitive behavioural programme for low back pain. The Back Skills Training (BeST) trial. Health Technol Assess. 2010 Aug;14(41):1-253, iii-iv. doi: 10.3310/hta14410. PMID 20807469
- [Background] Wiltsey Stirman S, Kimberly J, Cook N, Calloway A, Castro F, Charns M. The sustainability of new programs and innovations: a review of the empirical literature and recommendations for future research. Implement Sci. 2012 Mar 14;7:17. doi: 10.1186/1748-5908-7-17. PMID 22417162
- [Background] Hahne AJ, Ford JJ, Richards MC, Surkitt LD, Chan AYP, Slater SL, Taylor NF. Who Benefits Most From Individualized Physiotherapy or Advice for Low Back Disorders? A Preplanned Effect Modifier Analysis of a Randomized Controlled Trial. Spine (Phila Pa 1976). 2017 Nov 1;42(21):E1215-E1224. doi: 10.1097/BRS.0000000000002148. PMID 28263227
- [Derived] Fritz J, Almqvist L, Soderlund A, Wallin L, Sandborgh M. Patients' health outcomes after an implementation intervention targeting the physiotherapists' clinical behaviour. Arch Physiother. 2021 Oct 9;11(1):22. doi: 10.1186/s40945-021-00116-z. PMID 34625120